CLINICAL TRIAL: NCT04195581
Title: A Clinical Evaluation of Two Contact Lenses Used With Three Care Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C19-658 EX-MKTG-108
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Subjects will use each lens and solution combination for a month in random sequence for a total of six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (6):
- comfilcon A with Hy-Care Multi-purpose solution (Experimental): Subjects were randomized to wear each lens and solution combination for a month.
  Interventions: Device: comfilcon A
- comfilcon A with All in One Light Multi-purpose solution (Experimental): Subjects were randomized to wear each lens and solution combination for a month.
  Interventions: Device: comfilcon A
- comfilcon A with Refine One Step Hydrogen Peroxide Solution (Experimental): Subjects were randomized to wear each lens and solution combination for a month.
  Interventions: Device: comfilcon A
- fanfilcon A with Hy-Care Multi-purpose solution (Active Comparator): Subjects were randomized to wear each lens and solution combination for a month.
  Interventions: Device: fanfilcon A
- fanfilcon A with All in One Light multi-purpose solution (Active Comparator): Subjects were randomized to wear each lens and solution combination for a month.
  Interventions: Device: fanfilcon A
- fanfilcon A with Refine One Step Hydrogen Peroxide Solution (Active Comparator): Subjects were randomized to wear each lens and solution combination for a month.
  Interventions: Device: fanfilcon A

INTERVENTIONS:
Device: comfilcon A — Subjects were randomized to wear each lens and solution combination for a month.
  Arms: comfilcon A with All in One Light Multi-purpose solution; comfilcon A with Hy-Care Multi-purpose solution; comfilcon A with Refine One Step Hydrogen Peroxide Solution
Device: fanfilcon A — Subjects were randomized to wear each lens and solution combination for a month.
  Arms: fanfilcon A with All in One Light multi-purpose solution; fanfilcon A with Hy-Care Multi-purpose solution; fanfilcon A with Refine One Step Hydrogen Peroxide Solution

SUMMARY:
The objective of the study was to compare the clinical performance of the two contact lenses when used in combination with three care systems.

DETAILED DESCRIPTION:
This was a randomized, open-label, crossover study, controlled by cross-comparison. Subjects were randomized to wear each lens and solution combination for a month in random sequence; that is for a total of six months.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged 18-50 and have capacity to volunteer.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They are an existing wearer of reusable, single vision, spherical soft contact lenses.
5. They have a contact lens spherical prescription between -1.00 to - 6.50D (inclusive)
6. They have a spectacle cylindrical correction of -1.00D or less in each eye.
7. At dispensing, they can attain at least 0.20 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
8. They are willing to comply with the wear schedule (at least five days per week and for at least eight hours per day).
9. They agree not to participate in other clinical research for the duration of the study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They have had cataract surgery.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or breastfeeding.
8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
9. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
10. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, MCOptom FAAO FBCLA, Principal Investigator — Eurolens Research
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Subjects were randomized to wear each lens and lens solution combination for a month at random sequence for a total of 6 months.
  Contact lenses (comfilcon A, fanficon A) Lens Solution (Hy-Care, All in One Light and Refine One Step).
Period: Comfilcon A With All in One Light
Arm/Group | All Participants
Started | 28
Completed | 24
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Comfilcon A With Hy-Care
Arm/Group | All Participants
Started | 30
Completed | 25
Not Completed | 5
Not completed — Withdrawal by Subject | 5
Period: Comfilcon A With Refine One Step
Arm/Group | All Participants
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Fanfilcon A With All in One Light
Arm/Group | All Participants
Started | 28
Completed | 27
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Fanfilcon A With Hy-Care
Arm/Group | All Participants
Started | 28
Completed | 25
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Fanfilcon A With Refine One Step
Arm/Group | All Participants
Started | 29
Completed | 27
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to use each lens and solution combination for a month in random sequence; that is for a total of six months. Lenses (comfilcon A and fanfilcon A), Lens care solutions(Hy-Care, All in One Light and Refine One Step).
Arm/Group | Overall Study
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall Comfort will be assessed using vertical visual analogue scales (0-100) (0 - Causes Pain. Cannot be tolerated, 20 -Very uncomfortable, very irritating or annoying, 40 - Slightly uncomfortable, just irritating or annoying, 60 - Comfortable. Noticeable but not irritating, 80 - Very comfortable. Just felt occasionally, 100 - Excellent. Cannot be felt).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A With All in One Light Multi-purpose Solution: Subjects were randomized to wear comfilcon A with All in One Light Multi-purpose solution for a month.
- Comfilcon A With Hy-Care Multi-purpose Solution: Subjects were randomized to wear comfilcon A with Hy-Care Multi-purpose solution for a month.
- Comfilcon A With Refine One Step Hydrogen Peroxide Solution: Subjects were randomized to wear comfilcon A with Refine One Step Hydrogen Peroxide Solution for a month.
- Fanfilcon A With All in One Light Multi-purpose Solution: Subjects were randomized to wear fanfilcon A with All in One Light multi-purpose solution for a month.
- Fanfilcon A With Hy-Care Multi-purpose Solution: Subjects were randomized to wear fanfilcon A with Hy-Care Multi-purpose solution for a month.
- Fanfilcon A With Refine One Step Hydrogen Peroxide Solution: Subjects were randomized to wear fanfilcon A with Refine One Step Hydrogen Peroxide Solution for a month.
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 86.0 (12.0) | 81.6 (14.9) | 81.0 (17.1) | 87.7 (11.7) | 88.0 (9.5) | 82.7 (16.7)

2. Primary Outcome: Comfort on Insertion
Description: Comfort on insertion will be assessed using vertical visual analogue scales (0-100) (0 - Causes Pain. Cannot be tolerated, 20 -Very uncomfortable, very irritating or annoying, 40 - Slightly uncomfortable, just irritating or annoying, 60 - Comfortable. Noticeable but not irritating, 80 - Very comfortable. Just felt occasionally, 100 - Excellent. Cannot be felt).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 88.3 (12.7) | 85.8 (15.0) | 84.0 (17.1) | 88.6 (14.9) | 90.3 (10.6) | 87.3 (11.8)

3. Primary Outcome: Comfort Before Removal
Description: Comfort before removal will be assessed using vertical visual analogue scales (0-100) (0 - Causes Pain. Cannot be tolerated, 20 -Very uncomfortable, very irritating or annoying, 40 - Slightly uncomfortable, just irritating or annoying, 60 - Comfortable. Noticeable but not irritating, 80 - Very comfortable. Just felt occasionally, 100 - Excellent. Cannot be felt).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 80.0 (17.2) | 72.8 (17.8) | 74.2 (19.9) | 79.1 (17.2) | 82.4 (14.2) | 76.1 (19.9)

4. Secondary Outcome: Vision
Description: Vision will be assessed using vertical visual analogue scales (0-100) (0 - Unacceptable. Lens cannot be worn, 20 - Very poor. Marked and unacceptable reduction, 40 - Poor. Noticeable but acceptable reduction, 60 - Good. Occasional but acceptable reduction, 80 - Very good. Just noticeable and very occasional reduction, 100 -Excellent. Unaware of any visual loss)
Time Frame: One Month
Population: One subject was excluded from the analysis from fanfilcon A with All in One Light multipurpose solution and fanfilcon A with Refine One Step Hydrogen Peroxide Solution.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 26 | 25 | 26
units on a scale | 94.8 (7.7) | 91.4 (11.9) | 93.3 (9.3) | 90.9 (13.1) | 94.2 (7.7) | 93.4 (10.1)

5. Secondary Outcome: Variable Vision
Description: Variable Vision will be assessed using vertical visual analogue scales (0-100) (0 - Extremely poor. Intolerable levels of variation in vision, 20 - Very poor. Excessive variation in vision which definitely affects wearing my contact lenses, 40 - Poor. A level of variation in vision which is sometimes annoying, Good. Acceptable level of variation in vision, 80 - Very good. Very occasional or very slight sensation of variation in vision, 100 - Excellent. No variation in vision).
Time Frame: One Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 26 | 25 | 26
units on a scale | 92.5 (9.5) | 92.0 (11.5) | 91.8 (13.2) | 89.8 (15.4) | 92.8 (9.5) | 92.8 (10.9)

6. Secondary Outcome: Vision at Night
Description: Vision at night will be assessed using vertical visual analogue scales (0-100) (0 - Unacceptable. Lens cannot be worn, 20 - Very poor. Marked and unacceptable reduction, 40 - Poor. Noticeable but acceptable reduction, 60 - Good. Occasional but acceptable reduction, 80 - Very good. Just noticeable and very occasional reduction, 100 -Excellent. Unaware of any visual loss)
Time Frame: One Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 26 | 25 | 26
units on a scale | 92.5 (9.4) | 89.4 (13.8) | 91.6 (12.5) | 89.8 (13.0) | 91.3 (9.2) | 91.4 (11.0)

7. Secondary Outcome: Dryness
Description: Dryness will be assessed using vertical visual analogue scales (0-100) (0 - Extremely poor. Intolerable levels of dryness, 20 - Very poor. Dryness which definitely affects wearing my contact lenses, 40 - Poor. A level of dryness which is sometimes annoying, 60 - Good. Acceptable level of dryness, 80 - Very good. Very occasional or very slight sensation of dryness only, 100 - Excellent. I have no sensation of dryness whatsoever).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 85.5 (18.2) | 81.4 (17.4) | 81.5 (20.5) | 86.6 (11.3) | 86.3 (12.7) | 83.3 (16.3)

8. Secondary Outcome: Ocular Redness
Description: Ocular Redness will be assessed using vertical visual analogue scales (0-100) (0 - Extremely poor. Intolerable levels of redness, 20 - Very poor. Excessive redness which definitely affects wearing my contact lenses, 40 - Poor. A level of redness which is sometimes annoying, 60 - Good. Acceptable level of redness, 80 - Very good. Very occasional or very slight awareness of redness, 100 - Excellent. No redness).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 96.2 (8.6) | 92.6 (13.7) | 94.2 (10.9) | 95.8 (8.9) | 96.0 (5.6) | 92.7 (9.3)

9. Secondary Outcome: Burning/Stinging
Description: Burning/Stinging will be assessed using vertical visual analogue scales (0-100) (0 - Extremely poor. Intolerable levels of burning or stinging, 20 - Very poor. Excessive burning or stinging which definitely affects wearing my contact lenses, 40 - Poor. A level of burning or stinging which is sometimes annoying, 60 - Good. Acceptable level of burning or stinging, 80 - Very good. Very occasional or very slight sensation of burning or stinging, 100 - Excellent. No burning or stinging).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A With All in One Light Multi-purpose Solution: Subject were randomized to wear fanfilcon A with All in One Light multi-purpose solution for a month.
- Fanfilcon A With Hy-Care Multi-purpose Solution: Subject were randomized to wear fanfilcon A with Hy-Care Multi-purpose solution for a month.
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 93.4 (13.1) | 90.6 (14.7) | 85.7 (16.4) | 92.4 (14.3) | 95.7 (7.8) | 89.6 (14.8)

10. Secondary Outcome: Ease of Lens Insertion
Description: Ease of lens insertion will be assessed using vertical visual analogue scales 0-100. (0 - Unmanageable. Lenses impossible to insert, 20 - Very poor. Difficult and occasional unsuccessful insertion, 40 - Poor. Difficult with very occasional unsuccessful insertion, 60 - Good. Some problems but lens insertion usually successful, 80 - Very good. Occasional difficulty with lens insertion, 100 - Excellent. No problems with lens insertion).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 93.5 (9.0) | 91.2 (9.7) | 91.7 (12.4) | 91.6 (14.1) | 92.9 (9.7) | 91.3 (11.9)

11. Secondary Outcome: Ease of Lens Removal
Description: Ease of lens removal will be assessed using vertical visual analogue scales (0-100) ( 0 - Unmanageable. Lenses impossible to remove, 20 - Very poor. Difficult and occasional unsuccessful removal, 40 - Poor. Difficult with very occasional unsuccessful removal, 60 - Good. Some problems but lens removal usually successful, 80 - Very good. Occasional difficulty with lens removal, 100 - Excellent. No problems with lens removal).
Time Frame: One Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A With All in One Light Multi-purpose Solution: Subjects were randomized to wear comfilcon A with All in One Light Multipurpose solution for a month.
Arm/Group | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
Number analyzed (Participants) | 24 | 25 | 24 | 27 | 25 | 27
units on a scale | 92.1 (13.7) | 92.2 (12.6) | 91.6 (14.0) | 90.9 (10.7) | 92.0 (11.6) | 89.7 (12.5)

ADVERSE EVENTS:
Time Frame: Subjects were randomized to wear each lens and lens solution combination for a month at random sequence for a total of 6 months. Contact lenses (comfilcon A, fanficon A) Lens Solution (Hy-Care, All in One Light and Refine One Step).
Groups:
- Comfilcon A With Hy-Care Multi-purpose Solution: Subjects were randomized to wear comfilcon A with Hy-Care Multi-purpose solutionfor a month.
- Fanfilcon A With All in One Light Multi-purpose Solution: Subjects were randomized to wear fanfilcon A with All in One Light multi-purpose solutionfor a month.
- Fanfilcon A With Refine One Step Hydrogen Peroxide Solution: Subjects were randomized to wear fanfilcon A with Refine One Step Hydrogen Peroxide Solutionfor a month.
Arm/Group | Comfilcon A With Hy-Care Multi-purpose Solution | Comfilcon A With All in One Light Multi-purpose Solution | Comfilcon A With Refine One Step Hydrogen Peroxide Solution | Fanfilcon A With Hy-Care Multi-purpose Solution | Fanfilcon A With All in One Light Multi-purpose Solution | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/25 | 0/28 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/28 | 0/25 | 0/28 | 1/28 | 0/29
Other Adverse Events (participants affected / at risk) | 2/30 | 0/28 | 0/25 | 2/28 | 1/28 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comfilcon A With Hy-Care Multi-purpose Solution (N=30) | Comfilcon A With All in One Light Multi-purpose Solution (N=28) | Comfilcon A With Refine One Step Hydrogen Peroxide Solution (N=25) | Fanfilcon A With Hy-Care Multi-purpose Solution (N=28) | Fanfilcon A With All in One Light Multi-purpose Solution (N=28) | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution (N=29)
Corneal Infiltrate (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comfilcon A With Hy-Care Multi-purpose Solution (N=30) | Comfilcon A With All in One Light Multi-purpose Solution (N=28) | Comfilcon A With Refine One Step Hydrogen Peroxide Solution (N=25) | Fanfilcon A With Hy-Care Multi-purpose Solution (N=28) | Fanfilcon A With All in One Light Multi-purpose Solution (N=28) | Fanfilcon A With Refine One Step Hydrogen Peroxide Solution (N=29)
Corneal Infiltrate (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ocular Redness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04195581/Prot_SAP_000.pdf